CLINICAL TRIAL: NCT03924726
Title: Osseous Evidence Behind Micro-osteoperforation Technique in Accelerating Orthodontic Tooth Movement Towards Reducing Treatment Duration.
Brief Title: Osseous Evidence Behind Micro-osteoperforation in Accelerating Tooth Movement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, Wey Mang Chek, Assoc. Prof., University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FP018-2017A
Record Dates: First submitted 2019-04-12; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Orthodontics

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control and experimental (4 weeks MOP) (Other): This is a split mouth study. At the experimental site in group 1, three Micro-osteoperforation (MOP) were made directly at the buccal cortical bone of extracted first premolars sites, at equidistance from the canine and second premolar under local anaesthesia. This group received four sessions of MOPs at an interval of 4 weeks.
  Interventions: Procedure: Micro-osteoperforation (MOP)
- Control and experimental ( 8 weeks MOP) (Other): This is a split mouth study. This group received 2 sessions of Micro-osteoperforation (MOP) at an interval of 8 weeks.
  Interventions: Procedure: Micro-osteoperforation (MOP)
- Control and experimental (12 weeks MOP) (Other): This is a split mouth study. This group received 2 sessions of Micro-osteoperforation (MOP) at an interval of 12 weeks.
  Interventions: Procedure: Micro-osteoperforation (MOP)

INTERVENTIONS:
Procedure: Micro-osteoperforation (MOP) — Micro-osteoperforation technique is used to accelerate orthodontic tooth movement.

SUMMARY:
Introduction

The study aimed to investigate the effects of micro-osteoperforations (MOPs) on the changes in mandibular bone volume fraction (Bone Volume/Total Volume, BV/TV), in relation to the MOP effects on the rate of orthodontic tooth movement, using CBCT images. The other objective was to evaluate the effects of different frequency intervals (4 weeks, 8 weeks and 12 weeks) of MOPs on mandibular bone volume fraction (BV/TV), in relation to the rate of tooth movement.

Methods

In 24 participants, orthodontic force of 140-200 grams was applied for mandibular canine retraction. Three micro-osteoperforations (MOP's) were made according to the scheduled intervals of the three different groups (4, 8 and 12 weeks) directly at the mandibular buccal cortical bone of extracted first premolars sites. At the 12th week following MOP application, CBCT scans were performed. CT Analyser software was used to compute trabecular alveolar bone volume fraction (BV/TV).

DETAILED DESCRIPTION:
This study is a single centred, single-blinded, prospective randomised split-mouth clinical trial conducted at University of Malaya. The ethical approval for the present study was obtained from the institutional Medical Ethics Committee (DF CD1608/0059P). Written informed consents were obtained from all participants prior to the study. Cone beam computed tomography (CBCT) (Kodak 9000) images was used to assess the trabecular alveolar bone volume fraction (BV/TV) at micro-osteoperforations (MOPs) sides. The rate of orthodontic tooth movement was assessed by comparing the available space between control and MOP sites in three different interval groups. Twenty-four participants were selected according to the study selection criteria. Inclusion criteria was (1) aged 18 years and above at the start of the treatment, (2) molar relationship either Class I, < ½ unit Class II or Class III, (3) extraction of all four first premolar teeth as part of orthodontic treatment, (4) maximum anchorage required using mini-implant, (5) no systemic disease, (6) good oral hygiene and (7) no periodontal disease. Participants were excluded if they had significant vertical skeletal discrepancies, systemic diseases requiring long-term antibiotic use, phenytoin, cyclosporin, anti-inflammatory drugs, bisphosphonates, systemic corticosteroids or calcium channel blockers, poor oral hygiene for more than visits or active periodontal disease.

Sample size calculation

G*Power software (version 3.1.9.2) was used to calculate the total sample size of 24 using t tests to achieve a power of 80% and a level of significance of 5% (two sided), for detecting an effect size of 0.60 between pairs. However, 30 samples were selected to compensate for any dropouts during the study.

Demographic characteristic

Twenty-four participants were stratified in 3 study groups (4, 8 and 12 weeks) based on frequency intervention intervals. Ethnically, there were 11 Malay samples (45.8%), 10 Chinese samples (41.7%) and 3 Indian samples (12.5%). Gender and ethnic distribution was not equal within the study groups due to the limited sample size, as a result gender variance was not assessed in the present study.

Micro-osteoperforations and canine retraction

The lower dentition was bonded with preadjusted edgewise brackets (3M Unitek, 0.022" x 0.028" slot in MBT prescription), and the first and second molars banded (3M Unitek, 0.022" x 0.028" slot in MBT prescription). Mini-implants were inserted in the keratinised gingiva between the second premolars and first molars bilaterally for both indirect and direct anchorage purposes. Canine retraction was done one month after insertion of a stainless-steel working archwire (0.018 x 0.025-inch SS) (GAC PAK Stainless Steel ACCUFORM®), using power chain (3M Unitek Alastik TM elastomeric chain), with a force of 140-200 grams (measured directly using a Correx Force Tension gauge, Haag-Streit Diagnostics, Switzerland), engaged from the canines to the mini-implants. The distance of canine movement was recorded every four weeks with digital callipers accurate to 0.01 mm, for a period of 12 weeks.

Micro-osteoperforations were performed according to the scheduled intervals of the three different groups. At the experimental site, three micro-osteoperforations were made directly at the buccal cortical bone of extracted first premolars sites, at equidistance from the canine and second premolar under local anaesthesia. The MOPs were 2 mm apart in vertical direction and 3 mm depth. The first MOP were placed starting at the horizontal level of the cervical margin of the canine tooth and extending apically. Orlus Extra Thread mini-implant (1.6 mm width, 6 mm length) with a rubber stopper at a measured length (depth of micro-osteoperforation at 3 mm and soft tissue thickness was taken into consideration) was used to perform MOPs. Group1 received four sessions of MOPs, group 2 and group 3 received two sessions of MOPs. At the 12th week following MOP application, CBCT scans of the left and right mandibular quadrants (both control and intervention side) were acquired.

Radiographic evaluation of trabecular bone volume fraction

CBCT (Kodak 9000, Carestream) exposure parameters were 70KV, 8mA, 10.8s and voxel size of 76 µm. The DICOM® (Digital Imaging and Communications in Medicine) format of CBCT images were converted into BMP (Bitmap image) files using ImageJ software (Version 1.50i) before analysing the trabecular bone volume fraction (BV/TV) in CT Analyser software (version 1.11.0.0 copyright Sky Scan).

Blinding

Both the observers (orthodontic postgraduate students) were blinded to the frequency of MOP whilst analysing the bone volume fraction (BV/TV) using CT analyser software as CBCT files were labelled by random numbers.

Image Analysis

In CT Analyser, a region of interest (ROI) was identified between canine and second premolar teeth. The top slice of the ROI started from a slice apical to the cemento-enamel junction of canine. The bottom slice of the ROI was determined by subtracting 14.8mm from the Z-position of the upper slice on the axial view of CBCT image. A polygonal tool was used to mark the ROI at the top and bottom layers. Then a dynamic interpolation was applied to create an adaptive ROI. Then, the ROI was binarized using the threshold values obtained from the control side of each patient (Figure 4). The range of threshold values was determined by checking the threshold value of the cortical bone in the binary histogram. After binarization, the percentage of bone volume (BV/TV) was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above at the start of the treatment.
* Molar relationship either Class I, < ½ unit Class II or Class III.
* Extraction of all four first premolar teeth as part of orthodontic treatment.
* Maximum anchorage required using mini-implant.
* No systemic disease.
* Good oral hygiene.
* No periodontal disease.

Exclusion Criteria:

* Significant vertical skeletal discrepancies.
* Systemic diseases requiring long-term antibiotic use, phenytoin, cyclosporin, anti- inflammatory drugs, bisphosphonates, systemic corticosteroids or calcium channel blockers.
* Poor oral hygiene.
* Active periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of micro-osteoperforations (MOPs) on mandibular bone volume fraction (BV/TV). | 9 months
  BV/TV ratio was assessed between control and intervention sides to assess the effects of micro-osteoperforations (MOPs) on the changes in mandibular bone volume fraction (Bone Volume/Total Volume, BV/TV ).
To investigate the effects of micro-osteoperforations (MOPs) on the rate of orthodontic tooth movement. | 3 months
  The effect of MOPs on the rate of canine tooth movement was assessed by comparing the distance of canine retraction between control and micro-osteoperforations sides.

SECONDARY OUTCOMES:
The other objective was to evaluate the effects of different frequency intervals (4 weeks, 8 weeks and 12 weeks) of MOPs on mandibular bone volume fraction (BV/TV). | 9 months
  Bone volume fraction (BV/TV) was assessed by comparing the available space between control and MOP sites in three different interval groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wey M Chek, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.